CLINICAL TRIAL: NCT02728518
Title: Evaluation of the Safety and Efficacy of Nebulized Amikacin as Adjunctive Therapy in Hospital Acquired and Ventilator Associated Bacterial Pneumonia in Surgical Intensive Care Units
Brief Title: Nebulized Amikacin Versus Intravenous Amikacin in the Treatment of Nosocomial Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, NKhalek, Pharmacotherapy Specialist, National Heart Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHI-01
Record Dates: First submitted 2016-03-25; First posted 2016-04-05 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebulized Amikacin (Experimental): patients in this arm will take amikacin nebulizer 400 mg twice daily in addition to standard beta lactam
  Interventions: Drug: Nebulized Amikacin
- Amikacin Intravenous (Active Comparator): patients in this arm will take intravenous (IV) amikacin 20 mg/kg once daily in addition to standard beta lactam
  Interventions: Drug: Intravenous Amikacin

INTERVENTIONS:
Drug: Nebulized Amikacin — 400mg twice daily nebulized amikacin
  Arms: Nebulized Amikacin
Drug: Intravenous Amikacin — 20mg/kg once daily intravenous amikacin
  Arms: Amikacin Intravenous

SUMMARY:
The investigator's goal in this study is to evaluate the efficacy and safety of nebulized amikacin versus intravenous amikacin in patients with hospital and ventilator acquired pneumonia in surgical patients admitted to the intensive care units infected with gram negative bacilli

DETAILED DESCRIPTION:
prospective, randomized, controlled study on post-cardiac surgery patients , included two groups, over one year period. The first group was administered intravenous (IV) amikacin 20 mg/kg once daily. The second group was prescribed amikacin nebulizer 400 mg twice daily. Both groups were co-administered intravenous (IV) piperacillin/tazobactam empirically.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU
* Clinical suspicion of VAP or HAP defined by a new persistent radiological infiltrate and one of the following signs:
* purulent tracheal aspirations, or
* temperature of 38° or higher, or leucocyte count > 10000/ml or
* Positive culture sensitive to amikacin
* In case of empirical treatment, risk of multi resistant bacteria defined as follows:
* Antimicrobial therapy in preceding 90 days and
* Current hospitalization of 5 d or more

Exclusion Criteria:

* History of Asthma
* Multi organ failure or any psychiatric illness
* allergy to amikacin or intolerance to nebulized amikacin
* Myasthenia gravis.
* Severely impaired renal function (creatinine clearance lower than 10 mL/min or renal replacement therapy)
* Vestibulo-cochlear disease.
* Pregnancy.
* Brain death

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of cured patients in the nebulized amikacin group versus the proportion of cured patients in the intravenous group | through study completion, over one year

CONTACTS AND LOCATIONS:
Overall Officials: Nehal A Hassan, BCPS, Principal Investigator — National Heart Institute; Faten F El sayed, MD, Principal Investigator — National Heart Institute; Nirmeen A Sabry, Ph.D, Principal Investigator — Faculty of Pharmacy Cairo University

IPD SHARING:
Plan to Share IPD: Undecided